CLINICAL TRIAL: NCT04619199
Title: Influence of Socioeconomic and Environmental Factors on the Natural History of Idiopathic Pulmonary Fibrosis
Acronym: EXPOSOMFPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180343; 2019-A00825-52 (Other: ANSM - IDRCB)
Record Dates: First submitted 2020-10-23; First posted 2020-11-06 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Disease; Pulmonary Medicine
Keywords: socioeconomic Status; air pollution; Environmental exposure; Occupational exposure; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idiopathic Pulmonary Fibrosis (Experimental): Blood sample were performed during the study for all patients.
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample performed at the inclusion and during the follow-up.

SUMMARY:
Idiopathic Pulmonary Fibrosis(IPF) is the most common idiopathic interstitial lung disease whose cause is unknown. With age and gender, socio-economic factors are the most influential indicators of health. At present there is very little data on socio-economic factors in the IPF. The investigators hypothesize that a lower socio-economic level and / or exposure to various air pollutants may influence the IPF's natural history, including the severity of diagnosis and prognosis of the IPF. The investigators also hypothesize that the deleterious effect of air pollutants is modulated by individual susceptibility (shorter telomeres) and that this effect is related to oxidative stress and shortening of telomeres.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis is the most common idiopathic interstitial lung disease whose cause is unknown. However, it remains a rare disease, there is an incidence of approximately 4400 new patients per year in France. It is a serious disease with few therapeutic options and a median survival after diagnosis around 36 months. It is also responsible for high morbidity, with a marked deterioration in quality of life (dyspnea, cough, fatigue and anxiodepressive disorders) and significant functional impairment (respiratory failure) With age and gender, socio-economic factors are the most influential indicators of health. At present there is very little data on socio-economic factors in the IPF. The investigators hypothesize that a lower socio-economic level and / or exposure to various air pollutants may influence the IPF's natural history, including the severity of diagnosis and prognosis of the IPF. The investigators also hypothesize that the deleterious effect of air pollutants is modulated by individual susceptibility (shorter telomeres) and that this effect is related to oxidative stress and shortening of telomeres.

ELIGIBILITY:
Inclusion Criteria:

* Man woman over 18 years old
* Certain or probable Idiopathic Pulmonary Fibrosis determined by a multi-disciplinary discussion ("ATS / ERS / JRS / ALAT" 2018 criteria)
* Idiopathic Pulmonary Fibrosis with a diagnosis of less than 12 months
* Signed informed consent
* Patient affiliated to a social security scheme or universal health coverage or benefiting from state medical aid

Exclusion Criteria:

* Known cause of Diffuse Interstitial Lung Disease (including connectivity, Hypersensitivity pneumonitis or pneumoconiosis authenticated)
* Patient unable to answer questionnaires
* Pregnant or lactating woman
* Persons under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Determine if the household income is associated with the severity of the IPF at inclusion | Enrollment
  Patients will be classified into three groups: "lower" standard of living, "average" level and "higher" level. These groups are respectively defined by wages : less than 1000 euros, greater than or equal to 1000 euros and less than 4000 euros, and greater than or equal to 4000 euros.
  The severity of the IPF at baseline will be defined by the respiratory functional impact: a forced vital capacity (FVC) of less than 50% and / or a Carbon monoxide diffusion capacity of less than 30%.

SECONDARY OUTCOMES:
Describe the general and specific external environment of patients with IPF | Enrollment
  Collection of data on the general and specific external environment on patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution) on the severity of the IPF | Enrollment
  Collection of data about socio-economic and environmental factors, and about severity on patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution) on the quality of life | Enrollment
  Collection of data about socio-economic and environmental factors, and about quality of life on patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution) on the occurrence of an Acute Exacerbation | 24 months
  Collection of data about socio-economic and environmental factors, and about occurrence of an Acute Exacerbation on patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution) on the progress of the IPF | 24 months
  Collection of data about socio-economic and environmental factors, and about progression of IPF on patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution) on the mortality | 24 months
  Collection of data about socio-economic and environmental factors, and about mortality of patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution)on the existence and type of comorbidities | Enrollment
  Collection of data about socio-economic and environmental factors, and about existence and type of comorbidities on patients with IPF
Determine the impact of socio-economic factors and environmental factors (occupational domestic exposures and air pollution)on the diagnostic and management delay | Enrollment
  Collection of data about socio-economic and environmental factors, and about diagnostic and management delay on patients with IPF
Determine the impact of socio-economic factors and environmental factors on therapeutic decisions: anti-fibrotic treatments, access to transplantation | 24 months
  Collection of data about socio-economic and environmental factors (occupational domestic exposures and air pollution), and about therapeutic decisions (anti-fibrotic treatments, access to transplantation) on patients with IPF
Determine if the deleterious effect of air pollutants on the decline of respiratory function is dependent on the size of the telomeres | 24 months
  Collection of data about deleterious effect of air pollutants on the decline of respiratory function and about the length of telomers calculated with T/S ratio. Blood samples will be performed for analysis of biomarkers and oxidative stress in IPF, measurement of telomere length, MUC5B, TOLLIP and GSTT1 polymorphisms.

CONTACTS AND LOCATIONS:
Overall Officials: Lucile SESE, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Hilario NUNES, PHD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (16):
- France (16):
  - 001 - Service Pneumologie, Bobigny, Avicenne
  - 002 - Service Explorations Fonctionnelles Respiratoires, Bobigny, Avicenne
  - 003 - Service Pneumologie, Paris, Bichat
  - 016 - Service Pneumologie, Caen, CHU Caen Normandie
  - 010 - Service Pneumologie, Dijon, CHU Dijon
  - 013 - Service Pneumologie, Grenoble, CHU Grenoble
  - 008 - Service Pneumologie, Lille, CHU Lille
  - 015 - Service Pneumologie, Montpellier, CHU Montpellier
  - 007 - Service Pneumologie, Rennes, CHU Pontchaillou
  - 011 - Service Pneumologie, Strasbourg, CHU Strasbourg
  - 012 - Service Pneumologie, Tours, CHU Tours
  - 014 - Service Pneumologie, Meaux, GHEF
  - 005 - Service Pneumologie, Paris, HEGP
  - 006 - Service Pneumologie, Lyon, Hospices Civils de Lyon
  - 004 - Service de Pneumologie, Paris, Tenon
  - 009 - Service Pneumologie, Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duchemann B, Annesi-Maesano I, Jacobe de Naurois C, Sanyal S, Brillet PY, Brauner M, Kambouchner M, Huynh S, Naccache JM, Borie R, Piquet J, Mekinian A, Virally J, Uzunhan Y, Cadranel J, Crestani B, Fain O, Lhote F, Dhote R, Saidenberg-Kermanac'h N, Rosental PA, Valeyre D, Nunes H. Prevalence and incidence of interstitial lung diseases in a multi-ethnic county of Greater Paris. Eur Respir J. 2017 Aug 3;50(2):1602419. doi: 10.1183/13993003.02419-2016. Print 2017 Aug. PMID 28775045
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Raghu G, Rochwerg B, Zhang Y, Garcia CA, Azuma A, Behr J, Brozek JL, Collard HR, Cunningham W, Homma S, Johkoh T, Martinez FJ, Myers J, Protzko SL, Richeldi L, Rind D, Selman M, Theodore A, Wells AU, Hoogsteden H, Schunemann HJ; American Thoracic Society; European Respiratory society; Japanese Respiratory Society; Latin American Thoracic Association. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline: Treatment of Idiopathic Pulmonary Fibrosis. An Update of the 2011 Clinical Practice Guideline. Am J Respir Crit Care Med. 2015 Jul 15;192(2):e3-19. doi: 10.1164/rccm.201506-1063ST. PMID 26177183
- [Background] Cottin V. [French recommendations for idiopathic pulmonary fibrosis: An updated working document for clinicians]. Rev Mal Respir. 2017 Oct;34(8):789-790. doi: 10.1016/j.rmr.2017.09.005. No abstract available. French. PMID 29102032
- [Background] King TE Jr, Pardo A, Selman M. Idiopathic pulmonary fibrosis. Lancet. 2011 Dec 3;378(9807):1949-61. doi: 10.1016/S0140-6736(11)60052-4. Epub 2011 Jun 28. PMID 21719092
- [Background] Ley B, Collard HR, King TE Jr. Clinical course and prediction of survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2011 Feb 15;183(4):431-40. doi: 10.1164/rccm.201006-0894CI. Epub 2010 Oct 8. PMID 20935110
- [Background] Collard HR, Ryerson CJ, Corte TJ, Jenkins G, Kondoh Y, Lederer DJ, Lee JS, Maher TM, Wells AU, Antoniou KM, Behr J, Brown KK, Cottin V, Flaherty KR, Fukuoka J, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kolb M, Lynch DA, Myers JL, Raghu G, Richeldi L, Taniguchi H, Martinez FJ. Acute Exacerbation of Idiopathic Pulmonary Fibrosis. An International Working Group Report. Am J Respir Crit Care Med. 2016 Aug 1;194(3):265-75. doi: 10.1164/rccm.201604-0801CI. PMID 27299520
- [Background] Ley B, Ryerson CJ, Vittinghoff E, Ryu JH, Tomassetti S, Lee JS, Poletti V, Buccioli M, Elicker BM, Jones KD, King TE Jr, Collard HR. A multidimensional index and staging system for idiopathic pulmonary fibrosis. Ann Intern Med. 2012 May 15;156(10):684-91. doi: 10.7326/0003-4819-156-10-201205150-00004. PMID 22586007
- [Background] Raghu G, Amatto VC, Behr J, Stowasser S. Comorbidities in idiopathic pulmonary fibrosis patients: a systematic literature review. Eur Respir J. 2015 Oct;46(4):1113-30. doi: 10.1183/13993003.02316-2014. PMID 26424523
- [Background] Lantz PM, House JS, Lepkowski JM, Williams DR, Mero RP, Chen J. Socioeconomic factors, health behaviors, and mortality: results from a nationally representative prospective study of US adults. JAMA. 1998 Jun 3;279(21):1703-8. doi: 10.1001/jama.279.21.1703. PMID 9624022
- [Background] Gershon AS, Dolmage TE, Stephenson A, Jackson B. Chronic obstructive pulmonary disease and socioeconomic status: a systematic review. COPD. 2012 Jun;9(3):216-26. doi: 10.3109/15412555.2011.648030. Epub 2012 Apr 12. PMID 22497534
- [Background] Lederer DJ, Arcasoy SM, Barr RG, Wilt JS, Bagiella E, D'Ovidio F, Sonett JR, Kawut SM. Racial and ethnic disparities in idiopathic pulmonary fibrosis: A UNOS/OPTN database analysis. Am J Transplant. 2006 Oct;6(10):2436-42. doi: 10.1111/j.1600-6143.2006.01480.x. Epub 2006 Jul 26. PMID 16869805